CLINICAL TRIAL: NCT01009138
Title: Development and Evaluation of a Diabetes-specific Cognitive Behavioural Treatment (DS-CBT) for Diabetic Patients With Subthreshold Depression
Brief Title: Evaluation of a Diabetes-specific Cognitive Behavioural Treatment for Subthreshold Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Collaborators: German Diabetes Center (Other); University of Giessen (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, Prof. Dr., Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKZ 01GI0809
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Depressive Symptoms; Diabetes Mellitus
Keywords: Subthreshold Depression; Diabetes-related Distress; Minor Depression; Light affective Disorder; Subclinical depressive Symptoms; Diabetes mellitus; Late Complications; Markers of Inflammation
MeSH Terms: conditions — Depression; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes-Specific CBT (DS-CBT) (Experimental): Cognitive Behavioral Intervention (Group) focusing on Diabetes-Specific Problems
  Interventions: Behavioral: Diabetes-Specific CBT (DS-CBT)
- Standard Diabetes Education (Active Comparator): Standard Diabetes Education Lessons will be given to quantify the unspecific antidepressive Effects of Participation in Group Sessions with social Contact and Acquisition of Knowledge.
  Interventions: Behavioral: Standard Diabetes Education

INTERVENTIONS:
Behavioral: Diabetes-Specific CBT (DS-CBT) — 5 Group Sessions with a duration of 90 Minutes each, including the following cognitive-behavioral Intervention Methods focusing on Diabetes Distress and Hassles:
  * Problem Analysis and Definition
  * Problem Solving Intervention
  * Cognitive Restructuring
  * Activation of personal and social Resources
  * Goal Definition and Agreement
  Other Names: Diabetes-Specific Cognitive-Behavioral Group Sessions
  Arms: Diabetes-Specific CBT (DS-CBT)
Behavioral: Standard Diabetes Education — Standard Diabetes Education Lesson including
  * Health Care and specific Topics (e. g. Blood Pressure)
  * Social Aspects of Living with Diabetes
  * Diabetes Complications
  * Sports, Activities and Exercise
  * Healthy and unhealthy Food, Vitamins, Cooking Recommendations and Recipes
  * Foot Care: Exercises, Care and Control, Sensibility, Injuries, diabetic Neuropathy
  Other Names: Educative Group Lesson and Discussion
  Arms: Standard Diabetes Education

SUMMARY:
This work is supported by the "Kompetenznetz Diabetes mellitus (Competence Network for Diabetes mellitus)" funded by the Federal Ministry of Education and Research (FKZ 01GI0809).

Approximately one third of diabetic patients has elevated depressive symptoms. The majority of these patients are suffering from a subthreshold depression. In spite of the fact that subthreshold depression has an equivalent negative impact on the prognosis of diabetes as clinical depression, there is no specific intervention tool. The main objective of this project is to develop a diabetes specific cognitive behavioural treatment (DS-CBT) for diabetic patients with subthreshold depression. In a randomized trail DS-CBT is compared to standard diabetes education. A total of 188 diabetic patients will be recruited and randomly assigned to the two treatment conditions. The expected main outcome is the reduction of subthreshold depression under DS-CBT in a 12 month follow up. Secondary variables are improvement of glycaemic control, quality of life, diabetes self-management as well as reduction of health care costs and modification of inflammatory parameters.

DETAILED DESCRIPTION:
Elevated rates for depression in diabetic patients are of clinical significance for diabetology. Depressive disorders are doubled compared to patients without diabetes. A meta-analysis showed that a proportion of 20% of diabetic patients showed subthreshold depression, defined as elevated depressive symptoms without meeting criteria for clinical depression. Depression in diabetes is associated with a reduced quality of life, more diabetes related distress, and higher health related costs. But besides this, depression in diabetes seems to be an independent negative prognostic factor for morbidity and mortality. Furthermore subthreshold depression is a major barrier of an effective self-management of the disease.

Until now antidepressive therapies are only evaluated in clinically depressed diabetic patients. For the majority of depressed diabetic patients suffering from subthreshold depression no evaluated specific intervention concept exists. Since subthreshold depression often is associated with diabetes related distress a diabetes specific intervention was developed to support patients to increase their problem solving skills, modify their depressive cognitions and improve their coping with diabetes related distress. It consists of five sessions and is delivered as a group intervention.

This study is an efficacy trial. In this randomized trial the efficacy of this newly developed intervention is compared to a control condition consisting of five standard diabetes education lessons. The primary outcome variable is the reduction of depressive symptoms twelve months after the intervention. Secondary outcome variables are the quality of life, metabolic parameters, self-care behavior and other psychosocial aspects. Furthermore the possible covariation between change of depressive symptoms and inflammatory and immune markers will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Elevated depressive symptoms (regarding to CES-D)
* Age >= 18 and <=70
* Sufficient German language skills
* Informed consent

Exclusion Criteria:

* Current MDD
* Current schizophrenia/ psychotic disorder, eating disorder, bipolar disorder, addictive disorder, personality disorder
* Current antidepressive medication
* Current psychotherapy
* Severe physical illness (i.e. cancer)
* Being bedridden
* Guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Kulzer, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim e. V.; Norbert Hermanns, Prof., PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim e. V.; Thomas J Haak, Prof., MD, Study Director — Diabetes Zentrum Mergentheim; Forschungsinstitut der Diabetes Akademie Mergentheim e. V.
Locations (1):
- Forschungsinstitut der Diabetes Akademie Mergentheim e. V., Bad Mergentheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Tulu S, Telci Caklili O, Alkaya G, Oguz A. Comment on Hermanns et al. The Effect of a Diabetes-Specific Cognitive Behavioral Treatment Program (DIAMOS) for Patients With Diabetes and Subclinical Depression: Results of a Randomized Controlled Trial. Diabetes Care 2015;38:551-560. Diabetes Care. 2016 Jan;39(1):e12. doi: 10.2337/dc15-1692. No abstract available. PMID 26696661
- [Background] Hermanns N, Schmitt A, Reimer A, Ehrmann D, Haak T, Kulzer B. Response to Comment on Hermanns et al. The Effect of a Diabetes-Specific Cognitive Behavioral Treatment Program (DIAMOS) for Patients With Diabetes and Subclinical Depression: Results of a Randomized Controlled Trial. Diabetes Care 2015;38:551-560. Diabetes Care. 2016 Jan;39(1):e13-4. doi: 10.2337/dci15-0017. No abstract available. PMID 26696662
- [Result] Hermanns N, Schmitt A, Gahr A, Herder C, Nowotny B, Roden M, Ohmann C, Kruse J, Haak T, Kulzer B. The effect of a Diabetes-Specific Cognitive Behavioral Treatment Program (DIAMOS) for patients with diabetes and subclinical depression: results of a randomized controlled trial. Diabetes Care. 2015 Apr;38(4):551-60. doi: 10.2337/dc14-1416. Epub 2015 Jan 20. PMID 25605812
- [Result] Reimer A, Schmitt A, Ehrmann D, Kulzer B, Hermanns N. Reduction of diabetes-related distress predicts improved depressive symptoms: A secondary analysis of the DIAMOS study. PLoS One. 2017 Jul 10;12(7):e0181218. doi: 10.1371/journal.pone.0181218. eCollection 2017. PMID 28700718
- [Result] Schmitt A, Reimer A, Ehrmann D, Kulzer B, Haak T, Hermanns N. Reduction of depressive symptoms predicts improved glycaemic control: Secondary results from the DIAMOS study. J Diabetes Complications. 2017 Nov;31(11):1608-1613. doi: 10.1016/j.jdiacomp.2017.08.004. Epub 2017 Aug 9. PMID 28865713
- [Derived] Chernyak N, Kulzer B, Hermanns N, Schmitt A, Gahr A, Haak T, Kruse J, Ohmann C, Scheer M, Giani G, Icks A. Within-trial economic evaluation of diabetes-specific cognitive behaviour therapy in patients with type 2 diabetes and subthreshold depression. BMC Public Health. 2010 Oct 19;10:625. doi: 10.1186/1471-2458-10-625. PMID 20959009

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes-Specific CBT (DS-CBT): Cognitive Behavioral Intervention (Group) focusing on Diabetes-Specific Problems
  Diabetes-Specific CBT (DS-CBT): 5 Group Sessions with a duration of 90 Minutes each, including the following cognitive-behavioral Intervention Methods focusing on Diabetes Distress and Hassles:
  * Problem Analysis and Definition
  * Problem Solving Intervention
  * Cognitive Restructuring
  * Activation of personal and social Resources
  * Goal Definition and Agreement
- Standard Diabetes Education: Standard Diabetes Education Lessons with social Contact and Acquisition of Knowledge.
  Standard Diabetes Education: Standard Diabetes Education Lesson including
  * Health Care and specific Topics (e. g. Blood Pressure)
  * Social Aspects of Living with Diabetes
  * Diabetes Complications
  * Sports, Activities and Exercise
  * Healthy and unhealthy Food, Vitamins, Cooking Recommendations and Recipes
  * Foot Care: Exercises, Care and Control, Sensibility, Injuries, diabetic Neuropathy
Period: Overall Study
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Started | 106 | 108
Completed | 93 | 88
Not Completed | 13 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education | Total
Number analyzed (Participants) | 106 | 108 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15) | 43 (14) | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 121
  Male | 46 | 47 | 93
Type 1 diabetes [Number; unit: participants] | 63 | 78 | 141
Diabetes duration [Mean (Standard Deviation); unit: years] | 14 (10) | 14 (11) | 14 (11)
HbA1c (%-points) [Mean (Standard Deviation); unit: %-points] | 8.9 (1.8) | 8.9 (1.8) | 8.9 (1.8)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 30 (8) | 28 (6) | 29 (7)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms (CES-D Score)
Description: The Center for Epidemiologic Studies Depression Scale (CES-D) was used to assess depressive symptoms. The CES-D assesses the frequency of 20 typical symptoms of depression during the previous week on a 4-point Likert scale. Summing of the item scores estimates the total score with a range between 0 and 60 and higher scores indicating more severe depressive mood. Based on the measurement of depressive symptoms at baseline and 12-month follow up, the difference of the test scores between baseline and 12 month follow up was calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
Scores on a scale | -7.4 (11.4) | -2.7 (11.7)

2. Secondary Outcome: Quality of Life (EQ-5D TTO Score)
Description: The EuroQol Five Dimension Questionnaire (EQ-5D) was used to assess health-related quality of life (HRQOL). The EQ-5D assesses five dimensions of HRQOL using a 3-point scale. The item scores are weighted based on population data and used to calculate a standardised total score from 0 to 1 with higher scores indicating better HRQOL. Based on the measurement of HRQOL at baseline and 12-month follow up, the difference of the test scores between baseline and 12 month follow up was calculated.
Time Frame: Baseline,12 month FU
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
Scores on a scale | -0.01 (0.23) | -0.01 (0.25)

3. Secondary Outcome: Diabetes-specific Distress (PAID Score)
Description: The Problem areas in Diabetes Scale (PAID) was used to assess diabetes-specific distress. The PAID assesses diabetes-specific distress using 20 items and a five-point Likert scale (0 - 4). Item scores are summed and transformed to a range from 0 - 100 with higher scores indicating higher distress. Based on the measurement of diabetes-specific distress at baseline and 12-month follow up, the difference of the test scores between baseline and 12 month follow up was calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
Scores on a scale | -13.0 (18.9) | -4.2 (16.9)

4. Secondary Outcome: Diabetes Self-Care (SDSCA Score)
Description: The Summary of Diabetes Self-Care Activities Measure (SDSCA) was used to assess diabetes self-care. The SDSCA assesses the number of days of the previous week (0 - 7) on which several specific self-care activities (appropriate diet, physical activity, self-monitoring of blood glucose, foot care) were performed. The item scores are summed and averaged to a total score from 0 to 7 with higher scores indicating better overall self-care. Based on the measurement of diabetes self-care at baseline and 12-month follow up, the difference of the test scores between baseline and 12 month follow up was calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
Scores on a scale | -0.1 (1.1) | 0.0 (1.0)

5. Secondary Outcome: Diabetes Acceptance (AADQ Score)
Description: The Acceptance and Action Diabetes Questionnaire (AADQ) was used to assessment of diabetes acceptance. Using 11 items on diabetes-related experiential avoidance behaviours and a 5-point Likert response scale (1 - 5), the AADQ estimates the overall level of diabetes acceptance. Item scores are summed to a total score between 11 and 55 with higehr scores indicating better acceptance. Based on the measurement of diabetes acceptance at baseline and 12-month follow up, the difference of the test scores between baseline and 12 month follow up was calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
Scores on a scale | 2.5 (7.7) | 2.0 (6.6)

6. Secondary Outcome: Glycemic Control (HbA1c)
Description: The HbA1c was used as measure of glycemic control. All blood samples were analysed in a central laboratory using the Bio-Rad II Turbo analyser; the measurement units were %-points. Based on the measurement at baseline and 12-month follow up, the difference of the HbA1c values between baseline and 12 month follow up was calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (Standard Deviation); unit: %-points
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
%-points | -0.5 (2.0) | -0.7 (1.7)

7. Secondary Outcome: Inflammatory Marker IL-6
Description: The inflammatory marker Interleukin 6 (IL-6) was assessed as measure of distress-related immune activity. The differences of the serum-concentrations between baseline and 12 month follow up were calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
pg/ml | 0.0 [-0.6 to 0.4] | 0.1 [-0.6 to 0.5]

8. Secondary Outcome: Inflammatory Marker IL-1Ra
Description: The inflammatory marker Interleukin 1 receptor antagonist (IL-1Ra) was assessed as measure of distress-related immune activity. The differences of the serum-concentrations between baseline and 12 month follow up were calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
pg/ml | -100.5 [-261. to 28.8] | -70.8 [-171.8 to 11.8]

9. Secondary Outcome: Inflammatory Marker Hs-CRP
Description: The inflammatory marker high sensitivity C-reactive protein (hs-CRP) was assessed as measure of distress-related immune activity. The differences of the serum-concentrations between baseline and 12 month follow up were calculated.
Time Frame: Baseline, 12 month FU
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
mg/dl | 0.0 [-0.1 to 0.2] | 0.0 [-0.1 to 0.1]

10. Secondary Outcome: Health-care Costs: Health-care Utilisation
Description: Several aspects of interest regarding diabetes-related health-care costs were assessed in order to evaluate potential reductions of health-care costs following the treatment. Measurement was performed using retrospective interview refering to the previous 6 months: The assessed aspects were 1.) the number of out-patient medical appointments as a measure of costs related to health-care utilisation, 2.) the number of days on sick leave as a measure of costs related to non-productive time and 3.) the number of daily taken prescription medications as a measure of costs related to medication intake. For each aspect, the difference of the numbers between baseline and 12 month follow up was calculated.
Time Frame: Baseline, 12 months-FU
Measure: Mean (Standard Deviation); unit: number of medical appointment/half year
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
number of medical appointment/half year | -2.2 (15.4) | -1.4 (13.3)

11. Secondary Outcome: Health-care Costs: Non-productive Time
Description: as for outcome 10
Time Frame: Baseline, 12 months-FU
Measure: Mean (Standard Deviation); unit: number of days on sick leave/half year
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
number of days on sick leave/half year | -2.2 (33.2) | 5.8 (30.2)

12. Secondary Outcome: Health-care Costs: Medication Intake
Description: as for outcome 10
Time Frame: Baseline, 12 months-FU
Measure: Mean (Standard Deviation); unit: number of daily medications/half year
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Number analyzed (Participants) | 93 | 88
number of daily medications/half year | 0.7 (1.6) | 0.8 (2.0)

ADVERSE EVENTS:
Arm/Group | Diabetes-Specific CBT (DS-CBT) | Standard Diabetes Education
Serious Adverse Events (participants affected / at risk) | 11/106 | 21/108
Other Adverse Events (participants affected / at risk) | 28/106 | 28/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetes-Specific CBT (DS-CBT) (N=106) | Standard Diabetes Education (N=108)
Norwalk-Virus (Gastrointestinal disorders) | 3 | 4
Severe Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 7
Ketoacidosis (Metabolism and nutrition disorders) | 2 | 4
New diagnosis of diabetes long-term complication (General disorders) | 1 | 3
New diagnosis of cancer (General disorders) | 2 | 2
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetes-Specific CBT (DS-CBT) (N=106) | Standard Diabetes Education (N=108)
Nonsevere adverse event (General disorders) | 28 | 28 — Nonsevere adverse events were collected without regard to the specific Adverse Event Term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No